CLINICAL TRIAL: NCT04100174
Title: Focal HDR Brachytherapy Boost to Stereotactic Radiotherapy
Acronym: fBTsRT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18.295
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: focal brachytherapy boost to SBRT — As above

SUMMARY:
To determine if fBT+sRT is superior to standard care in terms of urinary toxicity by having fewer patients experience a minimal important decline (MID) in urinary irritation/obstructive QoL

DETAILED DESCRIPTION:
In this Phase IIR trial investigators primarily seek to determine if fBT boost (15Gy) to SBRT (35Gy/5) can be shown to be superior to standard care (whole-gland BT boost 15Gy to RT 37.5Gy/15) in terms of urinary toxicity by having fewer patients experience a minimal important decline (MID) in urinary irritation/obstructive QoL as measured by ePRO (EPIC-26) at 12 and 24 months post completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of prostate cancer planned for curative-intent HDR brachytherapy boost to external beam radiotherapy to the prostate gland.
* ECOG 0-1
* Charlson Comorbidity Index ≤ 4
* Imaging visible disease encompassing < 50% of the prostate gland and consistent with biopsy findings.

Exclusion - none

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Quality of Life | 12-24 months
  EPIC

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHUQ, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belliveau C, Barkati M, Delouya G, Taussky D, Beauchemin MC, Lambert C, Beaulieu L, Beliveau-Nadeau D, Nicolas B, Carrier JF, Vigneault E, Menard C. Focal HDR brachytherapy boost to stereotactic radiotherapy (fBTsRT) for prostate cancer: a phase II randomized controlled trial. Radiat Oncol. 2022 Dec 9;17(1):203. doi: 10.1186/s13014-022-02173-5. PMID 36494834